CLINICAL TRIAL: NCT03435510
Title: Implementation of the Live Donor Champion Program
Acronym: LDC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: IRB00161951
Record Dates: First submitted 2018-01-04; First posted 2018-02-19 (Actual); Last update posted 2025-12-22 (Actual); Status verified 2025-12

CONDITIONS: End-stage Renal Disease
Keywords: Live Donor Kidney Transplant; Education; Advocacy; Live Donor
MeSH Terms: conditions — Kidney Failure, Chronic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Live Donor Champion (Other): The Live Donor Champion program is the sole educational intervention for this trial. LDC consists of 6 monthly sessions of approx. 1 hour each. Each LDC session is led by a transplant physician or clinical coordinator. LDC sessions incorporate formal didactics, active-participant learning, personal stories, moderated group discussions, role-playing, and other skill-building exercises. LDC sessions are as follows: 1) education about ESRD, KT, and LDKT 2) communication skills building 3) Exploring social networks 4) sharing successful donor and recipient stories 5) encouraging candidate self-efficacy 6) Program Recap.
  Interventions: Behavioral: Live Donor Champion Program

INTERVENTIONS:
Behavioral: Live Donor Champion Program — Even with adequate education of live donation, many KT candidates still feel ill equipped to ask others to consider donating. Friends and family are often eager to help and may not be able to serve as donors themselves, but might be able to provide substantial instrumental support. An LDC is a friend or family member who serves as an advocate for the candidate in their pursuit of live donation. The Johns Hopkins Comprehensive Transplant Center has developed a 6-month program that provides education and advocacy training to waitlist candidates and their LDCs. The instrumental support provided by the LDC bridges a critical link between education and action.Using LDCs to increase live donation is a novel approach that has garnered widespread enthusiasm.
  Other Names: LDC Program

SUMMARY:
The Live Donor Champion Program is a clinical education program offered to patients placed on the waitlist for kidney transplantation at the Johns Hopkins Comprehensive Transplant Center. The goal of the program is to increase patient knowledge regarding end stage renal disease, kidney transplantation, and live kidney donation and to help patients identify potential live kidney donors. Patients are encouraged to bring family and friends to participate in the program and act as advocates on their behalf. These friends and family members are labeled "live donor champions" and work to assist the patient in spreading awareness about end stage renal disease, kidney transplantation, and live kidney donation.

The objectives of this project are to pilot-test and optimize strategies for the dissemination of the Live Donor Champion program in the clinical transplant center setting. The goals of the study are to develop an implementation protocol for centers who want to establish a live donor champion program at their institution.

DETAILED DESCRIPTION:
Live Donor Champion Concept: Even with adequate education of live donation, many kidney transplant candidates still feel ill equipped to ask others to consider donating. Friends and family are often eager to help and may not be able to serve as donors themselves, but might be able to provide substantial instrumental support. A "Live Donor Champion" (LDC) is a friend, family member, or community member who serves as an advocate for the candidate in their pursuit of live donation. The Johns Hopkins Comprehensive Transplant Center has developed a six-month program that provides education and advocacy training to waitlist candidates and their LDCs. The instrumental support provided by the LDC bridges a critical link between education and action. In pilot studies, candidates with an LDC were more likely to undergo Live Donor Kidney Transplant (LDKT) than matched controls. Using LDCs to increase live donation is a novel approach that has garnered widespread enthusiasm, including support from United Network for Organ Sharing.

Live Donor Champions (LDCs) as Instrumental Support for Transplant Candidates. Approaching potential donors is a daunting and overwhelming experience for Kidney Transplant (KT) candidates. Current educational programs address the medical aspects of dialysis, KT, and donation, but neglect the health communication skills to discuss transplantation and to spread awareness through their various social networks. While transplant candidates are hesitant to engage others in conversations about End Stage Renal Disease (ESRD) and live donation, friends, family members, or community members are eager to spread awareness and provide advocacy for the patient. In pilot studies, this intervention improved knowledge regarding LDKT and provided instrumental support to the transplant candidates. Understanding what factors are associated with the successful implementation of this program will enable its eventual dissemination at transplant centers nationwide ultimately improving nationwide education and awareness of LDKT. In order to successfully do so, a scientifically rigorous implementation study is necessary.

ELIGIBILITY:
Waitlist Candidates

Inclusion Criteria:

* Kidney transplant candidates aged≥18 added to the waitlist in the last year with no potential live donors are eligible.
* If there is an individual willing to donate, but the candidate is unwilling to consider this option or this particular individual, the candidate is eligible for the trial and may still benefit from identification of new donors or increased comfort accepting donation from others.
* Participants at University or University of Alabama must speak English. Participants at Northwestern University must speak English or Spanish.

Exclusion Criteria:

* Candidates with live donors currently under evaluation for donation will be excluded.
* Those with a previous kidney transplant will be excluded

Live Donor Champions Inclusion Criteria

* aged≥18
* English-speaking
* Be a "Live Donor Champion" (a friend, family member or community member willing to advocate for the wait-listed patient).

Exclusion Criteria

* <18, not English-speaking

LDC Administrators Inclusion Criteria

* aged≥18
* English-speaking
* Performed tasks related to implementing the LDC program

Exclusion Criteria

* <18, not English-speaking, and no affiliation with implementing the LDC program

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 111 (Actual)
Dates: Start 2018-05-30 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-04-30 (Actual)

PRIMARY OUTCOMES:
Acceptability - Implementation Outcome | within 2 years of enrollment
  Acceptability is the perception among implementation stakeholders that a given treatment, service, practice, or innovation is agreeable, palatable, or satisfactory. Acceptability will be measured qualitatively using an adapted Consolidated Framework for Implementation Research (CFIR) instrument. This instrument will be used during interviews with key stakeholders.
Adoption - Implementation Outcome | within 2 years of enrollment
  Adoption is defined as the intention or action to employ an innovation or practice. Adoption will be measured qualitatively using an adapted Consolidated Framework for Implementation Research (CFIR) instrument. This instrument will be used during interviews with key stakeholders.
Appropriateness - Implementation Outcome | within 2 years of enrollment
  Appropriateness is a qualitative measure of the perceived fit, relevance, or compatibility of the innovation for a given setting, provider, or consumer; and/or perceived fit of the innovation to address a particular issue. We will measure program appropriateness using an adapted Consolidated Framework for Implementation Research (CFIR) instrument. This instrument will be used during interviews with key stakeholders.
Cost - Implementation Outcome | within 2 years of enrollment
  Cost (incremental or implementation cost) is the cost impact of an implementation effort. Implementation cost will be assessed by estimations made during observational sessions of the intervention.
Feasibility - Implementation Outcome | within 2 years of enrollment
  Feasibility is defined as the extent to which a new treatment, or an innovation, can be successfully used or carried out within a given agency or setting. Feasibility will be assessed qualitatively using an adapted Consolidated Framework for Implementation Research (CFIR) instrument. This instrument will be used during interviews with key stakeholders.
Fidelity - Implementation Outcome | within 2 years of enrollment
  Fidelity is defined as the degree to which an intervention was implemented as prescribed in the original protocol or as it was intended by the developers. Fidelity will be qualitatively assessed using an adapted Consolidated Framework for Implementation Research (CFIR) instrument. This instrument will be used during interviews with key stakeholders.
Penetration - Implementation Outcome | within 2 years of enrollment
  Penetration is the integration of a practice within a setting or subsystem. Penetration of the LDC program within our two sites will be measured by calculating the number of eligible persons who use a service, divided by the total number of eligible.
Sustainability - Implementation Outcome | within 2 years of enrollment
  Sustainability is defined as the extent to which a newly implemented treatment is maintained or institutionalized within a service setting's ongoing, stable operations. Sustainability will be qualitatively assessed using an adapted Consolidated Framework for Implementation Research (CFIR) instrument. This instrument will be used during interviews with key stakeholders.

SECONDARY OUTCOMES:
Live donor kidney transplantation | within 1 year of enrollment
  Live donor kidney transplantation within one year of enrollment into the study will be collected/identified through electronic medical record system.
Live Donor Inquiries | within 1 year of enrollment
  Live Donor Inquiries on behalf of candidates will be collected/identified through electronic medical record system.
Knowledge of live donation and kidney transplantation | within 6 months of enrollment
  Knowledge of live donation of transplant candidates will be collected during the survey.
Comfort initiating conversations | within 6 months of enrollment
  Comfort initiating conversations with others about live donation will be collected during the survey.

CONTACTS AND LOCATIONS:
Overall Officials: Elizabeth King, MD PhD, Principal Investigator — Johns Hopkins University
Locations (2):
- United States (2):
  - Washington University in Saint Louis, St Louis, Missouri
  - University of Pennsylvania, Philadelphia, Pennsylvania

IPD SHARING:
Plan to Share IPD: No